CLINICAL TRIAL: NCT00659711
Title: The Effect of Januvia (Sitagliptin) on Oxidative Stress in Obese Type 2 Diabetic Subjects
Acronym: 1928
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Paresh Dandona, MD, Kaleida Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1931 Januvia
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Results first posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Januvia 100mg (Active Comparator): The first group will be started on 100 mg sitagliptin daily for 12 weeks
  Interventions: Drug: Januvia (Sitagliptin) 100 mg
- placebo (Placebo Comparator): will be placed on a placebo for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Januvia (Sitagliptin) 100 mg — The first group will be started on 100 mg sitagliptin daily for 12 weeks
  Other Names: januvia
  Arms: Januvia 100mg
Drug: Placebo — will be placed on a placebo for 12 weeks.
  Arms: placebo

SUMMARY:
Sitagliptin is a new oral hypoglycemic anti-diabetic drug used either alone or in combination with metformin or a thiazolidinedione for control of type 2 diabetes mellitus. Sitagliptin has been shown to have fewer side effects in the control of blood glucose values.

Obesity and diabetes are states of increased inflammation and can influence the free radicals and inflammatory markers (chemicals in the blood which increase due to inflammation in the body) and are also major risk factors for atherosclerotic disease. In this study we want to see the effect of sitagliptin on these markers. We believe that Sitagliptin may exert an anti-inflammatory effect in the human. The purpose of this study is to determine if the addition of sitagliptin to diabetic patients will provide added benefit. We believe that sitagliptin provides these added benefits by suppressing free radicals (charged substances that cause damage to the body) and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with age 20-75 years inclusive.
* Type 2 diabetes
* Males and Females BMI > 30
* Subjects on statins, ACE inhibitors, thiazolidenediones and antioxidants will be allowed as long as they are on stable doses of these compounds and the dosage in not changed during the course of study.
* BP under control -No change required to BP medications
* HbA1c > 7%

Exclusion Criteria:

* Coronary event or procedure (myocardial infarction, unstable angina, coronary artery bypass, surgery or coronary angioplasty) in the previous four weeks
* Pregnancy
* Hepatic disease (abnormal LFT's),Renal impairment (serum creatinine > 1.5),
* Participation in any other concurrent clinical trial
* Any other life-threatening, non-cardiac disease,
* Uncontrolled hypertension (BP > 160/100 mm of Hg)
* Congestive Heart Failure
* Use of an investigational agent or therapeutic regimen within 30 days of study
* Subjects on Exenatide, incretin or insulin therapy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Dandona, MD, Principal Investigator — Kaleida Health
Locations (1):
- 115 Flint Road, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Januvia 100mg | Placebo
Started | 12 | 10
Completed | 12 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Januvia 100mg | Placebo | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (4) | 53 (3) | 53.5 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 6 | 6 | 12
BMI [Mean (Standard Deviation); unit: kg/m^2] | 35 (1.5) | 35.4 (1.3) | 35.2 (1.4)
HbA1c [Mean (Standard Deviation); unit: percentage] | 7.6 (0.4) | 7.9 (0.3) | 7.7 (0.3)
Fasting glucose [Mean (Standard Deviation); unit: mg/dL] | 135 (13) | 148 (23) | 140 (18)

OUTCOME MEASURES:

1. Primary Outcome: Change in Reactive Oxygen Species (ROS) Generation by MNC, Protein and mRNA Expression of p47phox Subunit of NADPH Oxidase, in MNC's of Obese Type 2 Diabetic Patients
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Januvia 100mg | Placebo
Number analyzed (Participants) | 12 | 10
Percent change
  TNF-alpha | -39 (10) | 12 (8)
  TLR-4 | -23 (11) | 8 (5)
  TLR-2 | -35 (9) | 3 (5)
  JNK-1 | -19 (8) | 4 (7)
  IKK-beta | -17 (9) | 9 (8)
  CCR-2 | -24 (8) | 6 (4)

2. Secondary Outcome: Change in Oxidative Stress From Baseline to 12 Weeks
Description: To investigate that therapy with sitagliptin orally daily (100 mg) for 12 weeks decreases oxidized lipids (9-hydroxyoctadecadienoicacid (9-HODE) and 13-HODE) in plasma and F2-isoprostane in urine of obese type 2 diabetic patients
  Outcome measures given are calculated from the baseline - 12 weeks.
Time Frame: value at 12 weeks minus value at baseline
Measure: Mean (Standard Error); unit: mM
Arm/Group | Januvia 100mg | Placebo
Number analyzed (Participants) | 12 | 10
mM | -0.13 (0.06) | -0.06 (0.08)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: There were no participants at risk of an adverse event.
Arm/Group | Januvia 100mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes